CLINICAL TRIAL: NCT05271383
Title: Prospective Study to Evaluate the Performance (by the Assessment of Patient's Quality of Life) and the Safety of Global D's Implants of Cranio-maxillofacial Surgery Indicated for Orthognathic Surgery
Brief Title: Study Evaluating the Performance and Safety of Global D Implants Indicated for Orthognathic Surgery
Acronym: CMF-ORTHO
Status: Completed | Type: Observational
Sponsor: Global D (Industry)
Responsible Party: Sponsor
Other Study IDs: 2101-G-CMF-ORTHO-R
Record Dates: First submitted 2022-02-18; First posted 2022-03-09 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Orthognathic Surgery; Maxillofacial Abnormalities; Maxilla Fracture
Keywords: Orthognathic surgery; Performance; Security; Plates; Screw; Medical device; Cranio-maxillofacial
MeSH Terms: conditions — Maxillofacial Abnormalities; Maxillary Fractures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Male and female, major or minor, who will be treated by orthognathic surgery (maxillary, mandibular, maxillomandibular or/with genioplasty). The bone maturity of the participants (assessed by investigators) need to be sufficient for the treatment.
  Interventions: Device: Orthognathic surgery using Global D's implants.

INTERVENTIONS:
Device: Orthognathic surgery using Global D's implants. — Major or minor participants who will be treated by an orthognathic surgery with ORTRAUTEK® or MINITEK® implant(s).

SUMMARY:
This study is set up within the framework of the European Union regulation 2017/745 on medical devices. Its objective is to confirm the performance and safety of the Global D implants (ORTRAUTEK® and MINITEK®) used for orthognathic surgery.

DETAILED DESCRIPTION:
Study design : Non-interventional, prospective, multicentric, national, open-label, non-comparative study.

Investigators : 7 sites in France.

A statistical evaluation will be performed on those data in order to determine the performance and the security of those devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patient, major or minor, having reached bone maturity according to the judgement of the investigator,
* Patient having first orthognathic surgery (maxillary, mandibular, maxillomandibular or/with genioplasty)
* Patient who received orthodontic treatment prior to orthognathic surgery.
* Patient with abilities to read, understand and answer to the study quality of life questionnaire.
* Patient (and his legal representative if minor) who signed the study consent form.
* Patient affiliated to a social security system.

Exclusion Criteria:

* Patient allergic to one of the components of the implants
* Patient with physical or mental inabilities that will compromise the follow-up during the study
* Patient with acute or chronic infection (local or systemic)
* Person on legal protection
* Pregnant or breastfeeding women

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The study population is composed of male and female, major or minor, who will be treated by orthognatic surgery (maxillary, mandibular, maxillomandibular or/with genioplasty). The bone maturity of the participants (assessed by investigators) need to be sufficient for the treatment.
Sampling Method: Non-Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-08-02 (Actual)

PRIMARY OUTCOMES:
Performance of the Global D's implants used for orthognathic surgery, assessed by the Orthognathic Quality of Life Questionnaire (OQLQ) before and after the surgery. | 1 year
  The evolution of patient's quality of life will be assessed by comparing the score of the Orthognathic Quality of Life Questionnaire (OQLQ) before and after the surgery. The OQLQ can vary from 0 (better quality of life) to 88 (worst quality of life).

SECONDARY OUTCOMES:
Security of the Global D implants used for orthognathic surgery - Outcome Measure 1a | 6 weeks after the surgery
  Bone consolidation after the surgery, assessed by a correct dental occlusion on the postoperative image. This information is assessed 6 weeks after the surgery: correct occlusion (Yes/No).
Security of the Global D implants used for orthognathic surgery - Outcome Measure 1b | 6 weeks after the surgery
  Bone consolidation after the surgery, assessed by the alimentation of the patient. This information is assessed 6 weeks after the surgery: solid alimentation of the patient (Yes/No).
Security of the Global D implants used for orthognathic surgery - Outcome Measure 2 | 18 months
  Adverse events identification, assessment and follow-up.
Surgeon satisfaction on the implant's utilisation | Immediately following surgery
  Assessment by a satisfaction questionnaire, specially developed for the study, completed by the surgeon after the surgery. The surgeon evaluates each item using a likert scale (Highly Satisfied/ Satisfied/ Not very satisfied / Unsatisfied).

CONTACTS AND LOCATIONS:
Overall Officials: Pierre CORRE, MD, Principal Investigator — Cranio-maxillofacial surgeon
Locations (1):
- CHU de Nantes, Nantes, France